CLINICAL TRIAL: NCT03847402
Title: The Multi-site Study of the Early Integrated Intervention for Child Brain-developmental Disorders in China
Brief Title: The Early Integrated Intervention for Child Brain-developmental Disorders in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: National Key Research and Development Program of China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBDZXGY2018
Record Dates: First submitted 2019-02-11; First posted 2019-02-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-01

CONDITIONS: Brain Developmental Diseases; Autism Spectrum Disorder; Global Developmental Delay; Attention Deficit-Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GDD intervention (Experimental): The early integrated intervention for GDD
  Interventions: Behavioral: The early integrated intervention for GDD
- GDD non-intervention (Active Comparator): Community intervention for GDD
  Interventions: Behavioral: Community intervention for GDD
- ASD intervention (Experimental): The early integrated intervention for ASD
  Interventions: Behavioral: The early integrated intervention for ASD
- ASD non-intervention (Active Comparator): Community intervention for ASD
  Interventions: Behavioral: community intervention for ASD
- ADHD intervention (Experimental): The early integrated intervention for ADHD
  Interventions: Behavioral: The early integrated intervention for ADHD
- ADHD non-intervention (Active Comparator): Community intervention for ADHD
  Interventions: Behavioral: community intervention for ADHD

INTERVENTIONS:
Behavioral: The early integrated intervention for GDD — The early integrated intervention for GDD integrates developmental approaches with strategies of applied behavior analysis.
  Arms: GDD intervention
Behavioral: The early integrated intervention for ASD — The theoretical underpinnings of the early integrated intervention for ASD originate from Early Start Denver Model.
  Arms: ASD intervention
Behavioral: The early integrated intervention for ADHD — The methods of the early integrated intervention for ADHD includes behavior training, sensory integration training and psychological counseling
  Arms: ADHD intervention
Behavioral: community intervention for ASD — TEACCH (Treatment and Education of Autistic and related Communication- handicapped Children) intervention or ABA(applied behavior analysis) intervention
  Arms: ASD non-intervention
Behavioral: Community intervention for GDD — community intervention based on developmental approaches
  Arms: GDD non-intervention
Behavioral: community intervention for ADHD — School and family education
  Arms: ADHD non-intervention

SUMMARY:
This study is focused on developing the early integrated intervention for child brain-developmental disorders, including globe developmental delay (GDD), autism spectrum disorder (ASD), and attention deficit-hyperactivity disorder (ADHD), in China.

DETAILED DESCRIPTION:
The early integrated intervention of GDD and ASD is developed by Children's Hospital of Fudan University.

The early integrated intervention of ADHD is developed by Nanjing Brain Hospital.

ELIGIBILITY:
Inclusion Criteria:

* GDD: IQ<70, in more than 2 areas of development;
* ASD: Diagnose must meet the criteria of DSM-V;
* ADHD: Diagnose must meet the criteria of DSM-V, and IQ>70 tested by Wechsler Intelligence Scale；
* At least one of the parents could take part in the whole courses, and do the training at home.

Exclusion Criteria:

* Physical disability, visual or hearing loss;
* Combined other sever chronic diseases: liver or kidney function failure, rheumatic diseases, or tumor, and so on;

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline development quotient (DQ) in the Griffiths Development Scales-Chinese version at 1 year, 2 years for GDD and ASD | from enrollment to end of intervention (2 years). The DQ will be measured at the following time point: enrollment, 1 year, 2 years.
  Griffiths Development Scales-Chinese version consists of 5 subscales, which are locomotor scale, personal-social scale, eye& hand coordination scale, hearing& language scale. Each subscale has a development quotient. The developmental ages (DA) are referred from the norms and developmental quotients (DQ) are calculated by DA/CA (chronological age)*100. DQ for subscales have a mean of 100 (SD: 15). Higher DQ represent a better outcome. This is a repeate measurement
Change from baseline score of the Conners Early Childhood (Conners EC) at 1 year, 2 years for ADHD | from enrollment to end of intervention (2 years). The score of Conners EC will be measured at the following time point: enrollment, 1 year, 2 years.
  The Conners Early Childhood (Conners EC) aids in the early identification of behavioral, social, and emotional problems. It consists of 110 items. According to the 110 items of Conners EC, parents score children's behavioral frequency based on daily observations. The higher the score is, the more serious behavioral problems the children have. This is a repeate measurement

SECONDARY OUTCOMES:
Change from baseline score of the Communication and Symbolic Behavior Scales Developmental Profile-Infant Toddler Checklist（CSBS-DP-ITC）at 1 year, 2 years for ASD | from enrollment to end of intervention (2 years). The score of CSBS-DP-ITC will be measured at the following time point: enrollment, 1 year, 2 years.
  This is a parent-reported questionnaire widely used for screening communication disorders including ASD in infants and toddlers. The whole scale consists of 24 items divided into three subscales (social, speech, and symbolic composite) and an open question at the end. The changes in raw scores of each subscale and the whole scale partly reflect the change in social communication skills of children.This is a repeate measurement
Change from baseline intelligence quotient (IQ) in the Wechsler Intelligence Scale at 1 year, 2 years for ADHD | from enrollment to end of intervention (2 years). The IQ will be measured at the following time point: enrollment, 1 year, 2 years
  Wechsler Intelligence Scale consists of 2 subscales, which are verbal scale and performance scale. The intelligence quotient (IQ) are referred from the norms. Higher IQ represent a better outcome.This is a repeate measurement

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, MD, PhD, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan University, Shanghai, Shanghai Municipality, China